CLINICAL TRIAL: NCT05177796
Title: Enhancing Immunotherapy by Targeting the EGFR Pathway in Inflammatory Breast Cancer: A Phase II Study of Panitumumab (PmAb) and Pembrolizumab (Pembro) in Combination With Neoadjuvant Chemotherapy (NAC) in Patients With Newly Diagnosed Triple Negative Inflammatory Breast Cancer (TN-IBC)
Brief Title: Panitumumab and Pembrolizumab in Combination With Neoadjuvant Chemotherapy for the Treatment of Stage III-IV Triple Negative Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 participants recruited
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0715; NCI-2021-13704 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0715 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-12-14; First posted 2022-01-05 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-07

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Breast Inflammatory Carcinoma; Invasive Breast Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes; Panitumumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (panitumumab,pembrolizumab,neoajuvant chemotherapy) (Experimental): CYCLES 1-4: Patients receive pembrolizumab IV over 30 minutes and panitumumab IV over 30-60 minutes on day 1 of cycle 0. Cycle 0 continues for 7 days in the absence of disease progression or unacceptable toxicity. Patients then receive panitumumab IV over 30-60 minutes on days 1, 8, and 15 of cycles 1-3 and days 1 and 8 of cycle 4, pembrolizumab IV over 30 minutes on day 1 of cycles 2-4, paclitaxel IV over 1-3 hours on days 1, 8, and 15 of cycles 1-4, and carboplatin IV over 30 minutes on day 1, 8 and 15 of cycles 1-4. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  CYCLES 5-8: Patients receive standard of care treatment, including pembrolizumab IV over 30 minutes, doxorubicin IV over 15 minutes and cyclophosphamide IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Paclitaxel; Biological: Panitumumab; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; E7.6.3; Human IgG2K Monoclonal Antibody; MoAb ABX-EGF; MoAb E7.6.3; Monoclonal Antibody ABX-EGF; Monoclonal Antibody E7.6.3; Vectibix
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial tests whether panitumumab and pembrolizumab in combination with standard of care chemotherapy before surgery (neoadjuvant) works to shrink tumors in patients with stage III-IV triple negative breast cancer. Panitumumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as paclitaxel, carboplatin, doxorubicin, and cyclophosphamide work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving panitumumab and pembrolizumab in combination with neoadjuvant chemotherapy may kill more tumor cells in patients with triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the pathological complete response (pCR rate) of the proposed combination in patients with newly diagnosed triple-negative inflammatory breast cancer (TN-IBC).

SECONDARY OBJECTIVES I. To evaluate the surgical complication rate after the completion of the proposed treatment.

II. To determine the change of EGR1 related to the efficacy of proposed treatment. (Key Secondary Objective) III. To determine the immunological change of tumor microenvironment (TME) related to the efficacy of proposed treatment. (Key Secondary Objective) IV. To define the cutoff or threshold of changes of EGR1, which will correlate with the pCR.

V. To define the cutoff or threshold of immunological changes of TME, which will correlate with the pCR.

VI. To determine two-year recurrence-free survival (RFS) rates. VII. To determine two-year overall survival (OS) rates. VIII. To determine the safety and tolerability. IX. To determine the predictive biomarkers to predict the therapeutic response. (correlative study)

OUTLINE:

CYCLES 1-4: Patients receive pembrolizumab intravenously (IV) over 30 minutes and panitumumab IV over 30-60 minutes on day 1 of cycle 0. Cycle 0 continues for 7 days in the absence of disease progression or unacceptable toxicity. Patients then receive panitumumab IV over 30-60 minutes on days 1, 8, and 15 of cycles 1-3 and days 1 and 8 of cycle 4, pembrolizumab IV over 30 minutes on day 1 of cycles 2-4, paclitaxel IV over 1-3 hours on days 1, 8, and 15 of cycles 1-4, and carboplatin IV over 30 minutes on day 1, 8 and 15 of cycles 1-4. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 5-8: Patients receive standard of care treatment, including pembrolizumab IV over 30 minutes, doxorubicin IV over 15 minutes and cyclophosphamide IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, then every 6 months for 2 years from date of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to provide written informed consent for the trial
2. Female or male and >/= 18 years of age
3. Histological confirmation of invasive breast cancer. All histologic subtypes are eligible.
4. Clinical diagnosis of IBC and amenable to breast surgery Cohort 1 (safety run-in), stage III or de novo stage IV Cohort 2, stage III or de novo stage IV
5. Known ER, PR, and HER2 status defined as triple negative breast cancer (TNBC). TNBC is defined as ER and PR ≤ 10% by immunohistochemistry, and HER2 negative (defined as IHC 0, 1+, or 2+ and FISH negative. The positivity of FISH is determined as per ASCO/CAP guideline.(46)
6. ECOG performance status of 0-1.
7. Adequate organ function as determined by the following laboratory values:

   * ANC >/= 1,500/mcL
   * Platelets >/= 100,000/mcL
   * Hgb >/= 10g/dL
   * Creatinine levels <1.5 x ULN
   * Total bilirubin </= 1.5 x ULN,
   * ALT and AST </= 2.5 x ULN or </=5 x ULN for patients with liver metastases
8. Subjects of childbearing potential should be willing to use effective methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through at least 4 months after the last dose of study drug. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year. Effective methods of birth control include 1) Use of hormonal birth control methods: pills, shots/injections, implants (placed under the skin by a health care provider), or patches (placed on the skin); 2) Intrauterine devices (IUDs); 3) Using 2 barrier methods (each partner must use 1 barrier method) with a spermicide. Males must use the male condom (latex or other synthetic material) with spermicide. Females must choose either a Diaphragm with spermicide, or Cervical cap with spermicide, or a sponge (spermicide is already in the contraceptive sponge).
9. Negative serum or urine pregnancy test for subjects of childbearing potential.

Exclusion Criteria:

1. Any other previous or concurrent antitumor therapies for the current cancer diagnosis event.
2. Known diagnosis of immunodeficiency, which defined as on chronic systemic steroid therapy or any other forms of immunosuppressive therapy in excess of the equivalent of prednisolone 10 mg once daily.
3. History of malignancy (other than breast cancer) within 5 years, except basal cell carcinoma or squamous cell carcinoma of the skin, melanoma in-situ or in situ cervical cancer that has undergone potentially curative therapy.
4. Known active central nervous system metastases and/or carcinomatous meningitis.
5. Known significant cardiovascular disease, such as a history of myocardial infarction, acute coronary syndrome, Congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV, or history of CHF NYHA Class III or IV.
6. Ejection fraction < 50% by ECHO or MUGA.
7. Known active or uncontrolled autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids chronic corticosteroid use or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.

   History of (non-infectious) pneumonitis that required steroids or has a current diagnosis of pneumonitis.
8. An active infection requiring systemic therapy.
9. Gastrointestinal tract disease or defect or previous history of colitis or inflammatory bowel disease including Crohn's disease and ulcerative colitis.
10. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Known history of Human Immunodeficiency Virus.
12. Known active Hepatitis B or Hepatitis C
13. Received a live vaccine within 30 days before the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-07-26 (Estimated); Study Completion 2023-07-26 (Estimated)

PRIMARY OUTCOMES:
The ( pCR ) rate pathological complete response, defined as the absence of invasive carcinoma in the breast and the lymph nodes. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Nasrazad, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT05177796/ICF_000.pdf